CLINICAL TRIAL: NCT03547674
Title: Tuned Versus Untuned Ankle-foot Orthoses in Children and Adolescents With Cerebral palsy_AFO-Study
Brief Title: Tuned Versus Untuned Ankle-foot Orthoses in Children and Adolescents With Cerebral Palsy
Acronym: AFO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2018-00541; ks17Rutz3 (Other: CTU Basel)
Record Dates: First submitted 2018-05-17; First posted 2018-06-06 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Community Health Workers; Shoes

STUDY DESIGN:
Intervention Model Description: Prospective, cross-sectional within-subjects comparison
Masking Description: Gait analysis under 4 conditions (barefoot, shoes only, untuned AFO with shoes, tuned AFO with shoes) will be performed in a random order: To determine the order, the 4 conditions will be noted on a piece of paper and randomly picked from an envelope.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- barefoot (Active Comparator): Gait analysis under 4 conditions (barefoot, shoes only, untuned AFO with shoes, tuned AFO with shoes) will be performed in a random order.
  Interventions: Other: barefoot
- shoes only (Active Comparator): Gait analysis under 4 conditions (barefoot, shoes only, untuned AFO with shoes, tuned AFO with shoes) will be performed in a random order.
  Interventions: Other: shoes only
- untuned AFO with shoes (Active Comparator): Gait analysis under 4 conditions (barefoot, shoes only, untuned AFO with shoes, tuned AFO with shoes) will be performed in a random order.
  Interventions: Other: untuned AFO with shoes
- tuned AFO with shoes (Experimental): Gait analysis under 4 conditions (barefoot, shoes only, untuned AFO with shoes, tuned AFO with shoes) will be performed in a random order.
  Interventions: Other: tuned AFO with shoes

INTERVENTIONS:
Other: barefoot — Gait analysis under 4 conditions (barefoot, shoes only, untuned AFO with shoes, tuned AFO with shoes) will be performed in a random order.
  Arms: barefoot
Other: shoes only — Gait analysis under 4 conditions (barefoot, shoes only, untuned AFO with shoes, tuned AFO with shoes) will be performed in a random order.
  Arms: shoes only
Other: untuned AFO with shoes — Gait analysis under 4 conditions (barefoot, shoes only, untuned AFO with shoes, tuned AFO with shoes) will be performed in a random order. AFO are walking aids to improve gait pathologies. They are custom-built using plaster casts. AFO for equinus and/or drop foot pathologies are specifically indicated to control excessive ankle plantar flexion. Push-up elements that return the energy from the stance-phase to support lifting the foot during the swing-phase (similar to a spring) are used.
  Arms: untuned AFO with shoes
Other: tuned AFO with shoes — Gait analysis under 4 conditions (barefoot, shoes only, untuned AFO with shoes, tuned AFO with shoes) will be performed in a random order. Modular AFO tuning means that patients try different pushup elements with varying stiffness and design before the final design is determined.
  Arms: tuned AFO with shoes

SUMMARY:
Cerebral palsy (CP) in children and adolescents is frequently accompanied by gait abnormalities. Ankle-foot orthoses (AFO) have been suggested to improve the gait pattern. Compared to conventional AFO, modular AFO offer the opportunity to tune its response to the patient's gait characteristics and/or functional maturity. However, the evidence level is still small and AFO tuning is not yet established in clinical routine. The study will investigate individual tuning of custom-built ankle-foot-orthoses (AFO) using gait analyses

ELIGIBILITY:
Inclusion Criteria:

* Patients in outpatient treatment from the University Children's Hospital Basel (UKBB)
* Informed Consent provided as documented by signature
* Confirmed diagnosis of cerebral palsy
* Confirmed diagnosis of spastic equinus and/ or drop foot,
* Gait pathologies treated with conventional AFO
* Gross Motor Function Classification System (GMFCS) level I or II

Exclusion Criteria:

* Other neuromuscular diseases
* Previous surgical treatment to improve gait pathologies
* Injections of Botulinum toxin 6 month prior to study inclusion
* Inability or unwillingness to follow the procedures of the gait analysis

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
gait profile score (GPS) | at end of study, an average of 1 month
  overall score calculated from all kinematic parameters (joint rotation angles) of the affected leg and expressed as the deviation from the normal gait cycle in degrees. The mean GPS was anticipated to be 9° with standard deviation of 1.4° [2]. A good (r = 0.5) correlation of GPS for the within-subjects comparison was assumed. The non-inferiority margin was set at the minimally clinically important difference of 1.6°.

SECONDARY OUTCOMES:
Movement analysis profile (MAP) | at end of study, an average of 1 month
  calculated from kinematic parameters and expressed as the deviation from the normal gait cycle in degrees. The MAP consists of individual scores for each joint rotation angle (pelvic tilt, pelvic obliquity, pelvic rotation, hip flexion/extension, hip abduction/adduction, hip rotation, knee flexion/extension, ankle dorsiflexion/extension and foot progression) of the affected leg
spatio-temporal parameter | at end of study, an average of 1 month
  calculated from kinematic parameters and expressed as the deviation from the normal gait cycle in degrees,Spatio-temporal parameters are walking speed (m/s), cadence (steps/min x 100) and stride length (m) of the affected leg

CONTACTS AND LOCATIONS:
Overall Officials: Erich Rutz, PD MD, Principal Investigator — Universitäts-Kinderspital beider Basel (UKBB)
Locations (1):
- University of Basel Children's Hospital (UKBB), Basel, Switzerland

REFERENCES:
- [Result] Schroder JH, Barandun GA, Leimer P, Morand R, Gopfert B, Rutz E. Novel Modular Walking Orthosis (MOWA) for Powerful Correction of Gait Deviations in Subjects with a Neurological Disease. Children (Basel). 2023 Dec 26;11(1):30. doi: 10.3390/children11010030. PMID 38255343